CLINICAL TRIAL: NCT03784144
Title: Effect of the Cognitive Strategy During Trunk Muscle Endurance in Patients With Lumbar Hernia Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital San José, Chile (Other)
Collaborators: Hospital Clínico La Florida (Other)
Responsible Party: Principal Investigator, Carlos Cruz Montecinos, Principal Investigator, Hospital San José, Chile
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: HSanJose
Record Dates: First submitted 2018-12-19; First posted 2018-12-21 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Low Back Pain; Disk Herniated Lumbar
Keywords: Muscle endurance; Biering-Sorensen Test; Prone Plank Test.; Dual task; time to failure
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Each test will be assessed in different days following a randomized order.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Strategy (Experimental): Performing a mathematical subtracting task (starting at 300, by sevens)
  Interventions: Diagnostic Test: Biering-Sorensen Test and Prone Plank Test
- Control (Active Comparator): The patients will perform both tests without any cognitive condition
  Interventions: Diagnostic Test: Biering-Sorensen Test and Prone Plank Test

INTERVENTIONS:
Diagnostic Test: Biering-Sorensen Test and Prone Plank Test — All patients will be encouraged to achieve the maximum time to task failure, stopped only by muscular fatigue or pain precluding to maintain the position.

SUMMARY:
Muscle endurance will be evaluated on two exercises: Biering-Sorensen Test and Prone Plank Test. Each test will be assessed in different days following a randomized order.

DETAILED DESCRIPTION:
All patients will be encouraged to achieve the maximum time to task failure, stopped only by muscular fatigue or pain precluding to maintain the position. Each exercise will perform under two conditions.

On the control condition, the patients will perform both tests without any cognitive condition, while on the experimental condition they will be instructed to perform both tests while performing a mathematical subtracting task (starting at 300, by sevens).

The starting condition will be randomly assigned with a 5-minute rest prior to the next condition. Time to task failure and pain perception using a visual analog scale will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-50 years.
* Surgery of lumbar discectomy or lumbar arthrodesis with at least 3 months of evolution.
* Acceptance to participate in the study.

Exclusion Criteria:

* History of previous surgery in the lower extremities.
* Recent trauma (<6 months).
* Use of corticosteroids.
* Pregnancy.
* Cauda equina syndrome.
* Marrow-level lesions.
* Progressive neurological involvement.
* History of rheumatological diseases.
* Inability to perform the test measurement.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 15 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-01-07 (Actual); Study Completion 2019-01-22 (Actual)

PRIMARY OUTCOMES:
Time to task failure | through study completion, an average of 2 week
  Time in seconds from 0 to failure, where higher values represent a best muscle endurance.
Pain evaluation | through study completion, an average of 2 week
  Pain will be measured by the Visual Analog Scale for pain (VAS) from 0 to 10, where higher values represent a worse outcome.

SECONDARY OUTCOMES:
Pain Interference: Kinesiophobia | through study completion, an average of 2 week
  Kinesiophobia will be evaluated by Tampa Scale for Kinesiophobia (TSK-11SV) (Spanish adaptation. Gómez-Pérez, López-Martínez y Ruiz-Párraga, 2011). Scoring: Items are summed, with a total score from 11-44 and higher values represent a worse outcome (more pain interference in behavior).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico La Florida, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No
Muscle endurance will be evaluated on two exercises: Biering-Sorensen Test and Prone Plank Test.

REFERENCES:
- [Background] Gomez-Perez L, Lopez-Martinez AE, Ruiz-Parraga GT. Psychometric Properties of the Spanish Version of the Tampa Scale for Kinesiophobia (TSK). J Pain. 2011 Apr;12(4):425-35. doi: 10.1016/j.jpain.2010.08.004. PMID 20926355
- [Derived] Cruz-Montecinos C, Nunez-Cortes R, Guzman-Gonzalez B, Andersen LL, Garcia-Masso X, Calatayud J. The Relevance of Dual Tasking for Improving Trunk Muscle Endurance After Back Surgery. Arch Phys Med Rehabil. 2021 Mar;102(3):463-469. doi: 10.1016/j.apmr.2020.07.015. Epub 2020 Sep 2. PMID 32888906